CLINICAL TRIAL: NCT00943540
Title: Pharmacokinetic and Safety Pilotstudy of RAltegravir and Atazanavir in a Once DAily Dose Regimen in HIV-1 Infected Patients (PRADA)
Brief Title: Pharmacokinetic and Safety Study of Raltegravir and Atazanavir in a Once Daily Dose Regimen in HIV-1 Infected Patients
Acronym: PRADA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: D.M. Burger, PhD, PharmD, Radboud University Medical Centre Nijmegen
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCN-AKF 08.07
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: HIV Infection; HIV Infections
Keywords: pharmacokinetics; single dose; raltegravir; Treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — Atazanavir Sulfate; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Raltegravir BID-QD (Experimental): Week 1-4
  * 600 mg of atazanavir to be taken once daily
  * 400 mg of raltegravir to be taken twice daily
  * 300 mg of lamivudine (or 200 mg of emtricitabine) to be taken once daily
  Week 5-8
  * 600 mg of atazanavir to be taken once daily
  * 800 mg of raltegravir to be taken once daily
  * 300 mg of lamivudine (or 200 mg of emtricitabine) to be taken once daily
  Interventions: Drug: raltegravir QD; Drug: atazanavir; Drug: lamivudine (or emtricitabine)

INTERVENTIONS:
Drug: raltegravir QD — Raltegravir 800mg QD
Drug: atazanavir — atazanavir
Drug: lamivudine (or emtricitabine) — lamivudine (or emtricitabine)

SUMMARY:
The licensed dose of raltegravir is 400 mg twice daily with or without food. Raltegravir is metabolized predominantly through glucuronidation by UGT1A1. Atazanavir increases the plasma concentrations of raltegravir 400 mg twice daily by 72% due to inhibition of UGT 1A1.

This suggests that combined use of atazanavir and a lower dose frequency of raltegravir, once daily for example, is possible. Another reason why raltegravir most likely can be applied is that its pharmacodynamic effect is not related to Cmin but to AUC which is expected to be similar for an 800mg QD dose when compared to 400mg BD. Phase III clinical trials evaluating QD dosing of raltegravir are currently ongoing and interim results are expected to be published in mid 2009.

A regimen of atazanavir and raltegravir in combination with lamivudine or emtricitabine may be a well tolerated and effective NNRTI-, and ritonavir-sparing regimen that could be an attractive option for both first and second line (after NRTI/NNRTI failure) treatment regimens.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected as documented by positive HIV antibody test and confirmed by Western Blot.
* Subject is at least 18 years of age at the day of screening.
* Subject is able and willing to sign the Informed Consent Form prior to screening evaluations.
* HIV-1 RNA < 40 copies/mL for at least 6 months on antiretroviral therapy.
* Subject has no history of previous virological failure or documented resistance mutations

Exclusion Criteria:

* History of sensitivity/idiosyncrasy to the drug or chemically related compounds or excipients, which may be employed in the trial.
* Relevant history or current condition that might interfere with drug absorption, distribution, metabolism or excretion.
* Inability to understand the nature and extent of the trial and the procedures required.
* Pregnant female (as confirmed by an HCG test performed less than 3 weeks before the first dose) or breast-feeding female.
* Abnormal serum transaminases determined as levels being > 5 times upper limit of normal (see Appendix A for normal ranges of clinical laboratory values).
* Concomitant use of medications that interfere with raltegravir or atazanavir pharmacokinetics: rifampicin, irinotecan, midazolam, triazolam, ergotamine, dihydroergotamine, cisapride, pimozide, lovastatin, simvastatin, indinavir, proton pump inhibitors, H2 receptor antagonists, St. john's wort, Ginkgo Biloba, didanosine, tenofovir, efavirenz, nevirapine, antacids, clarithromycin, phenytoin, phenobarbital, carbamazepine.
* Active hepatobiliary or hepatic disease (including chronic hepatitis B infection).
* Alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
pharmacokinetics of raltegravir | after two weeks of reference treatment and after two weeks of test treatment

SECONDARY OUTCOMES:
Viral load | after two weeks treatment with the reference treatment and after two weeks treatment with the test treatment
Adverse events | entire trial

CONTACTS AND LOCATIONS:
Overall Officials: David Burger, Principal Investigator — Radboud University Medical Center
Locations (4):
- University of Bonn, Bonn, Germany
- Netherlands (3):
  - Rijnstate Hospital Arnhem, Arnhem
  - Radboud University Medical Centre Nijmegen, Nijmegen
  - Erasmus Medical Center Rotterdam, Rotterdam

REFERENCES:
- [Result] Jansen A, Colbers EP, van der Ven AJ, Richter C, Rockstroh JK, Wasmuth JC, van Luin M, Burger DM. Pharmacokinetics of the combination raltegravir/atazanavir in HIV-1-infected patients. HIV Med. 2013 Aug;14(7):449-52. doi: 10.1111/hiv.12029. Epub 2013 Mar 18. PMID 23506243